CLINICAL TRIAL: NCT01524861
Title: Sympathetic Heart Innervation in Patients With Previous Experience of Transient Stress-induced Cardiomyopathy (Tako-Tsubo): Effects of α-lipoic Acid and L-acetyl Carnitine Therapies.
Brief Title: Sympathetic Heart Innervation in Patients With Tako-Tsubo Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, Assistant Professor of Internal Medicine, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IT 278354
Record Dates: First submitted 2012-01-23; First posted 2012-02-02 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Apical Ballooning Syndrome; Nervous System Diseases, Sympathetic
Keywords: Tako-Tsubo; Sympathetic heart innervation; MIBG; Alpha-lipoic acid; L-acetyl carnitine
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Autonomic Nervous System Diseases | interventions — Thioctic Acid; Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 30 subjects receive placebo (placebo group)
  Interventions: Drug: Placebo
- alpha-lipoic acid (Experimental): 30 subjects receive alpha-lipoic acid, 400 mg/day per os bis in die (800 mg/day)(ALA group)
  Interventions: Drug: alpha-lipoic acid
- L-acetil-carnitine (Experimental): 30 subjects receive L-acetyl carnitine, 500 mg per os bis in die (1000 mg/day) (LAC group)
  Interventions: Drug: L-acetyl carnitine

INTERVENTIONS:
Drug: Placebo — a placebo tablet bis in die for 12 months
  Arms: Placebo
Drug: alpha-lipoic acid — alpha-lipoic, tablets of acid 400 mg bis in die (800 mg/day), for 12 months
  Arms: alpha-lipoic acid
Drug: L-acetyl carnitine — L-acetyl carnitine tablets, 500 mg bis in die (1000 mg/day), for 12 months
  Arms: L-acetil-carnitine

SUMMARY:
Stress (tako-tsubo) cardiomyopathy (SC) is a rapidly reversible form of acute heart failure reported to be triggered by stressful events and associated with a distinctive left ventricular (LV) contraction pattern.

SC mimics acute coronary syndrome and is accompanied by reversible left ventricular apical ballooning in the absence of angiographically significant coronary artery stenosis. sympathetic activity dysfunction appears to play a very important role in the pathophysiology of takotsubo cardiomyopathy.

In most cases, myocardial scintillography with 123Imetaiodobenzylguanidine (MIBG) showed altered captation of the radiotracer in several heart segments. In particular, the apical myocardium has poor sympathetic innervations and an uptake reduction in MIBG tracer.

A hypothesis for this finding could be that the intense discharge of adrenalin, acting on heart segment with different and abnormal innervation, may produce a transient heart failure characterized by a particular shape of the left ventricle.

While studies have shown that heterogeneous MIBG distribution, decreased MIBG uptake and increased norepinephrine content were completely prevented by α-lipoic acid or by L-acetyl carnitine administrations in diabetic cardiomyopathy, no studies have examined the effects of these therapies on tako-tsubo cardiomyopathy.

On this basis, the investigators study will evaluate whether the dysfunction of adrenergic cardiac innervation, evaluated by MIBG, persist after previous experience of transient stress-induced cardiac dysfunction. Moreover, the investigators will assess whether the medications that restore sympatho-vagal alterations in diabetic cardiomyopathy, such as α-lipoic acid and L-acetyl carnitine, will improve the adrenergic cardiac innervation, in patients with SC.

DETAILED DESCRIPTION:
Study design Each patient will be assessed with history and physical examination, 12-lead ECG, serum troponin, coronary arteriography, and LV angiogram (an average of 6 hours after admission to the hospital), with echocardiography and 123Imetaiodobenzylguanidine (MIBG) myocardial scintillography. All patients were admitted to the cardiac care unit after coronary angiography. Currently recommended treatments for acute coronary syndromes (ACS), with therapy directed at relieving myocardial ischemia and preventing thrombotic complications, were provided to all patients. For each patient, the Charlson score index, 8 which represents the most studied and evaluated comorbidity index, will be calculated. At discharge, surviving patients with established SC will be managed and followed for 12 month after the event, as outpatients. At discharge, the surviving patients will be randomly assigned to alpha-lipoic acid 800 mg/day treatment (ALA group), or L-acetyl carnitine 1000 mg/day treatment (LAC group) or placebo (control group). With regard to the full medical therapy, the protocol stated that the use of concomitant treatment should be uniform, between the groups, and according to evidence-based international guidelines for ACS in all patients. Following discharge, patients were asked to return to our outpatient clinic for follow-up evaluation at 6 and 12 months after the initial event of SC.

Coronary Angiography Coronary angiograms at baseline, immediately after percutaneous coronary intervention (PCI) will be performed in at least 2 orthogonal views after intracoronary nitroglycerin. The analyses of all angiographic data will be performed by operators who were unaware of the study groups (Toshiba, Infinix CS-i).

Echocardiography LV function will be evaluated in all patients by two-dimensional echocardiography at admission, 6 and 12 months after the discharge.

MIBG imaging. MIBG imaging will be performed in all patients shortly after admission and at 6 and 12 months after the discharge. MIBG will be performed with a The standard protocol for 123I-MIBG cardiac imaging requires that drugs that interfere with 123I-MIBG uptake be withheld. A comprehensive listing of prescription and over-the-counter drugs that interfere with 123I-MIBG biodistribution, and the time for which they should be withheld, has been published . Thyroid uptake of unbound 123I is blocked with 500 mg of potassium perchlorate given orally 30 min before 123I-MIBG injection. Between 148 MBq and 370 MBq of 123I-MIBG are injected intravenously at rest. Both planar and SPECT images are acquired 15 min after injection (early) and 4 h after injection (delayed). A dual head gammacamera (ECAM Siemens, Erlangen - Germany) equipped with a low-energy - high resolution collimator was used. A 20% window is usually centered over the 159-keV photopeak of 123I for imaging. Anterior planar images of the chest are acquired using a 256 x 256 matrix. single photon emission computed tomography (SPECT) images are acquired using a 64 x 64 matrix over 180°, from the right anterior oblique position to the left posterior oblique position. Planar imaging allows for global assessment of cardiac innervation, whereas SPECT allows for regional evaluation. Quantitative evaluations will be performed with a standard protocol previously described.

ELIGIBILITY:
Inclusion Criteria:

* acute onset of a cardiovascular event, usually associated with substernal chest pain, initially regarded as ST-segment elevation myocardial infarction/evolving coronary syndrome;
* systolic dysfunction, predominantly characterized by akinesia/hypokinesia of the mid-to-distal portion of the LV chamber, with hypercontractile basal LV;

Exclusion Criteria:

* presence, by angiography, of significant atherosclerotic luminal narrowing in each of the 3 epicardial coronary arteries (0 to < 25%) (- presence of pheochromocytoma, myocarditis, or hypertrophic cardiomyopathy.
* coexisting conditions that limited life expectancy to less than 12 months or that could affect a patient's compliance with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Adrenergic cardiac innervation at 6 and 12 months | 0, 6 and 12 months
  The improvement of adrenergic cardiac innervation as determined by quantitative MIBG

SECONDARY OUTCOMES:
Change from Baseline in the markers of inflammation at 6 and 12 months | 0, 6 and 12 months
  Serum concentrations of IL-6 and IL-18 will be determined using a highly sensitive, quantitative sandwich enzyme assay. High-sensitivity TNF-α will assayed by immune-nephelometry. CRP will be determined using automated turbidimetry.
Change from Baseline in the markers of oxidative stress at 6 and 12 months | 0, 6 and 12 months
  Nitrotyrosine plasma concentration, will be assayed by enzyme-linked immunosorbent assay.
Change from Baseline in the markers of myocardial damage at 6 and 12 months | 0, 6 and 12 months
  Serum levels of Troponin I, miR-1, miR-133a, and miR-499 will be evaluated.
Change from Baseline in the markers of sympathetic tone at 6 and 12 months | 0, 6 and 12 months
  Plasma levels of catecholamines and their metabolites will measured by HPLC; brain natriuretic peptide and neuropeptide Y will be measured by enzyme immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli; Raffaele Marfella, MD, PhD, Principal Investigator — Dept Geriatric and Metabolic diseases SUN, Naples, Italy
Locations (1):
- Dept Geriatric and Metabolic diseases SUN, Naples, Italy